CLINICAL TRIAL: NCT06407687
Title: Comparative Effects of Electro Dry Needling Versus Dry Needling on Pain, Endurance and Range of Motion in Patients With of Quadratus Lumborum Syndrome
Brief Title: Compare Electrodry Needlig and Dry Needling in Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0183
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Quadratus Lumborum Syndrome
Keywords: Dry Needling; Endurance; pain; range of motion; Quadratus Lumborum Syndrome
MeSH Terms: conditions — Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric dry needling (Experimental): Group A will receive Electrical Dry Needling along with conventional physiotherapy. The parameters for Electro dry needling will be needles of 30×0.25 mm, 50×0.25 mm sizes Frequency 80-100 Hz, Duration 10-30 minutes and intensity as tolerated.
  Interventions: Device: Electro Dry Needlig
- Dry needling (Active Comparator): Group B will receive Dry Needling along with conventional Physiotherapy in which parameters will be dry needles will be 30×0.25 and 50×0.25 mm sizes.
  Interventions: Device: dry needling

INTERVENTIONS:
Device: Electro Dry Needlig — Electro Dry Needling is a modified form of dry needling which utilises an electro-stimulation unit connected via cables to fine filament needles. The combination of dry needling with electro-stimulation often prolongs the pain relief effect by blocking nerve pathways and preventing pain signals from travelling to the brain.
  Arms: Electric dry needling
Device: dry needling — Dry needling is a technique that acupuncturists, physical therapists and other trained healthcare providers use to treat musculoskeletal pain and movement issues.
  Arms: Dry needling

SUMMARY:
Mechanical low back pain (LBP) generally results from an acute traumatic event, but it may also be caused by cumulative trauma. The severity of an acute traumatic event varies widely, from twisting one's back to being involved in a motor vehicle collision. Mechanical LBP due to cumulative trauma tends to occur more commonly in the workplace and Quadratus Lumborum injury plays an important role in causing MLBP. The aim of this study is To compare the effects of Electrical Dry Needling and Dry Needling on pain, endurance and range of motion in patients with Quadratus Lumborum Syndrome.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Ali Afzal Shah Dispensary and Inam ul Haq Clinic Lahore through consecutive sampling technique on 40 patients which will be allocated using simple random sampling and patients will be divided in Group A and B. Group A will receive Electrical Dry Needling along with conventional physiotherapy. The parameters for Electro dry needling will be needles of 30×0.25 mm, 50×0.25 mm sizes Frequency 80-100 Hz, Duration 10-30 minutes and intensity as tolerated 1 session per week along with 5 day conventional physiotherapy a week for 4 weeks. Group 2 will receive Dry Needling along with conventional Physiotherapy in which parameters will be dry needles will be 30×0.25 and 50×0.25 mm sizes once per week and 5 days of conventional Physiotherapy per week for 4 weeks. Data will be analyzed during SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 45 years.
* Male and females both included.
* Muscle hypersensitivity on palpation
* Deep aching pain in sides of the lower back.
* Positive side-bridge test (Right < 83.2 sec and Left < 81.5 sec)
* Positive Simon's criteria for Quadratus Lumborum
* Patients with NPRS <7
* ODI score of < 40
* Decreased Lumber Side flexion and extension ROM
* Positive apperent Leg Length Discrepancy with more than 2 cm
* Negative Laslet's criteria for sacroiliac dysfunction

Exclusion Criteria:

* People with real leg length discrepancy
* People with any other medical condition Including Lumbar fracture, Spondylolisthesis, Ankylosing Spondylysis, Rheumatoid Arthritis. All these conditions will be ruled out with carefully history and examination.
* People taking any other form of treatment including corticosteroids, non-steroidal anti-inflammatory drugs or analgesics.
* People with previous history of surgical treatment for Lumbar spine. o People with neurological deficits or systemic illness

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 4th week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Leg length Discrepancy | 4th week
  Involves measuring limb length with a tape measure between 2 defined points, in the stand. Two common points are the anterior iliac spine and the medial malleolus or the anterior inferior iliac spine and lateral malleolus
Endurance | 4th week
  The McGill Torso Endurance Tests are a useful battery of tests that assess all sides of the trunk allowing us to assess the endurance capacity of the torso muscles or if there is an imbalance between these three muscle groups which can contribute to low-back dysfunction and core instability.
Range of motion | 4th week
  Universal goniometer will be used to measure side binding ROM of Lumber Spine in atient with Quadratus Lumborum Syndrome.Universal goniometer is tool that has two arms and a fulcrum in which one arm remains fixed and the other arm moves to measure the ROM. The norm side bending ROM of Lumber Spine is 20 degress on each side. Its reliability is 0.97 and validity is 0.98
Disability | 4th week
  ODI scoring is used to measure the disability of the patient. ODI score system consists of sections which includes a score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. And in this study the patients with moderate disability will be included for the study and its Reliability is 0.88 and validity is 0.93

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Ali Afzal Shah Dispensary, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borenstein D. Mechanical low back pain--a rheumatologist's view. Nat Rev Rheumatol. 2013 Nov;9(11):643-53. doi: 10.1038/nrrheum.2013.133. Epub 2013 Sep 10. PMID 24018549
- [Background] Trompeter K, Fett D, Platen P. Prevalence of Back Pain in Sports: A Systematic Review of the Literature. Sports Med. 2017 Jun;47(6):1183-1207. doi: 10.1007/s40279-016-0645-3. PMID 28035587
- [Background] Wong AYL, Karppinen J, Samartzis D. Low back pain in older adults: risk factors, management options and future directions. Scoliosis Spinal Disord. 2017 Apr 18;12:14. doi: 10.1186/s13013-017-0121-3. eCollection 2017. PMID 28435906
- [Background] Pandey E, Kumar N, Das SJPOTJ. Effect of stretching on shortened quadratus lumborum muscle in non specific low back pain. 2018;11(2):80-6.
- [Background] Will JS, Bury DC, Miller JA. Mechanical Low Back Pain. Am Fam Physician. 2018 Oct 1;98(7):421-428. PMID 30252425
- [Background] MHMD H, Choudhury M, Mojumder M. A COMPARATIVE STUDY OF TREATMENT OF CHRONIC BACKACHE BETWEEN CONVENTIONAL METHOD AND TRIGGER POINT INJECTIONS (TPI).
- [Background] Bryner P, HSR GD. Unilaterol bock poin: ci cose series of quodroitus lumborum. 1996.
- [Background] Grover C, Christoffersen K, Clark L, Close R, Layhe S. Atraumatic Back Pain Due to Quadratus Lumborum Spasm Treated by Physical Therapy with Manual Trigger Point Therapy in the Emergency Department. Clin Pract Cases Emerg Med. 2019 May 29;3(3):259-261. doi: 10.5811/cpcem.2019.4.42788. eCollection 2019 Aug. PMID 31404175
- [Background] Fernández-de-las-Peñas C, Dommerholt JJTpdnae, approach c-b. Basic concepts of myofascial trigger points (TrPs). 2013:3-19.
- [Background] de Franca GG, Levine LJ. The quadratus lumborum and low back pain. J Manipulative Physiol Ther. 1991 Feb;14(2):142-9. PMID 1826922